CLINICAL TRIAL: NCT03480906
Title: An Evaluation of the Usability and Patient Tolerability for Microtherapeutic Dosing of Commercially Available Ocular Medication Via the Eyenovia Microdose Delivery System (MiDD)
Brief Title: Eyenovia MiDD Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eyenovia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: EYN-POC-PG-21
Record Dates: First submitted 2018-03-13; First posted 2018-03-29 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Intraocular Pressure
MeSH Terms: interventions — Latanoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microdose administration (Experimental): Latanoprost ophthalmic solution administered as a microdose using the Eyenovia MiDD
  Interventions: Drug: Latanoprost
- Eyedrop administration (Active Comparator): Latanoprost ophthalmic solution administered as an eyedrop
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: Latanoprost — Latanoprost ophthalmic solution administered as a microdose spray
  Arms: Microdose administration
Drug: Latanoprost — Latanoprost ophthalmic solution administered as an eyedrop
  Arms: Eyedrop administration

SUMMARY:
This study is to evaluate the usability and patient tolerability for microtherapeutic dosing of commercially available ocular medication via the Eyenovia microdose delivery system (MiDD)

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients without significant ocular pathology and mean unmedicated diurnal intraocular pressure (IOP) in the range of of 17-27 mmHg
* Willing to forego use of contact lenses during study period
* Presence of cognition an dexterity necessary to follow MiDD drug administration instructions
* Female subjects must be 1-year postmenopausal, surgically sterilized, or if of childbearing potential, have a negative serum pregnancy test

Exclusion Criteria:

* Prior clinically significant ocular history or abnormal eye exam
* Use of ocular medication within 30 days of screening
* Use of oral steroid within 30 days of screening, or anticipated need for ocular steroid treatment during study period
* History of drug or alcohol abuse within 1 year of screening
* Lid squeezer
* Presence of disabling arthritis or limited motor coordination that would limit self-handling of the MiDD
* Participation in any interventional study of an investigational drug or device within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-03-17 (Actual); Study Completion 2018-03-17 (Actual)

PRIMARY OUTCOMES:
Successful microtherapeutic administration to the ocular surface | Treatment Day 3
  Cumulative percent of cases in which microdose medication is delivered to the ocular surface as evaluated by the treating physician and an independent observer

CONTACTS AND LOCATIONS:
Overall Officials: Reuben Orillac, MD, Principal Investigator — Clinica de Ojos Orillac-Calvo; Ernesto Calvo, MD, Principal Investigator — Clinica de Ojos Orillac-Calvo
Locations (1):
- Clinica de Ojos Orillac-Calvo, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No